CLINICAL TRIAL: NCT03877523
Title: Effects of Cocarnit on Macrophages Polarization in Type 2 Diabetic Patients
Brief Title: Cocarnit Effects on Macrophages Polarization
Acronym: COMP-DM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute for Atherosclerosis Research, Russia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IAR-CS1
Record Dates: First submitted 2019-03-11; First posted 2019-03-15 (Actual); Last update posted 2019-03-21 (Actual); Status verified 2019-03

CONDITIONS: Diabetes Mellitus, Type 2; Diabetes Complications
Keywords: Cocarnit; Diabetes Mellitus; Macrophages polarization
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Complications; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cocarnit (Experimental): disodium adenosine triphosphate trihydrate 10mg, cocarboxylase 50mg, cyanocobalamin 500mg and nicotinamide 20mg
  Interventions: Dietary Supplement: Cocarnit

INTERVENTIONS:
Dietary Supplement: Cocarnit — a metabolic complex

SUMMARY:
Cocarnit is a metabolic complex containing disodium adenosine triphosphate trihydrate, cocarboxylase, cyanocobalamin and nicotinamide.

Aim: To test the effects of Cocarnit on pro- and anti-inflammatory activation of blood-derived monocytes-macrophages from Type 2 diabetic patients.

Study design: Measurements of stimulated and basal secretion of TNF-alpha and CCl-18 before and at 2 and 4 hours after single intramuscular administration of Cocarnit at first day and after 30 days of follow-up in 40 Type 2 diabetic patients with/without polyneuropathy.

Methods: The profile of monocyte polarization was determined in vitro in primary cell culture of blood-derived monocytes-macrophages after pro-inflammatory stimulation by bacterial lipopolysaccharide and after anti-inflammatory stimulation by interleukin-4, according to tumor necrosis factor (TNF) and CCL18 chemokine secretion, respectively.

DETAILED DESCRIPTION:
Diabetes mellitus (DM) is the most common endocrine disease, and its social significance is associated with early disability and high mortality. Indicators of diabetes mellitus decompensation are its chronic complications, the most common one is a diabetic polyneuropathy. In recent years a large number of papers demonstrate the role of the chronic inflammatory process in the development of type 2 DM. Macrophages play a key role in the development of the inflammatory response. Macrophages are the main cells producing pro-inflammatory cytokines, which cause a cascade of reactions leading to the development of insulin resistance, that is the important factor of the pathogenesis of type 2 DM. There are two main types of activation of macrophages under the influence of T-helper cells 1 and 2. The first type is classical activation of macrophages that is a response to pro-inflammatory stimuli, such as interferon-gamma or lipopolysaccharide. Classically activated macrophages are well studied and characterized by the secretion of reactive oxygen species and pro-inflammatory cytokines such as TNF-alpha, interleukins 1,6,12. The second type is alternative activation of macrophages that is the result of the influence of anti-inflammatory cytokines, such as interleukins 4,10,13 or anti-inflammatory mediators, for example, glucocorticoids. The result of alternative activation of macrophages is the expression of anti-inflammatory cytokines such as antagonist receptor interleukin 1, interleukin 10, CCL18, haptoglobin receptor CD163, scavenger receptor type1.

Cocarnit is a metabolic complex containing disodium adenosine triphosphate trihydrate 10mg, cocarboxylase 50mg, cyanocobalamin 500mg and nicotinamide 20mg.

The aim of the present study is to test the effects of Cocarnit on pro- and anti-inflammatory activation of blood-derived monocytes-macrophages from Type 2 diabetic patients.

The profile of monocyte polarization was determined in vitro in primary cell culture of blood-derived monocytes-macrophages after pro-inflammatory stimulation by bacterial lipopolysaccharide and after anti-inflammatory stimulation by interleukin-4, according to tumor necrosis factor (TNF) and CCL18 chemokine secretion, respectively.

Study design: Open label study included 40 Type 2 diabetic patients divided into two groups:

1. Newly-diagnosed type-2 DM - 20 participants;
2. Type-2 DM with polyneuropathy - 20 participants.

The following measurements are held:

1. stimulated and basal secretion of TNF-alpha before and at 2 and 4 hours after single intramuscular administration of Cocarnit at first day and 30 days of follow-up.
2. stimulated and basal secretion of CCl-18 before and at 2 and 4 hours after single intramuscular administration of Cocarnit at first day and after 30 days of follow-up.

The research database is compiled upon completion of the study and then a statistical analysis of the results is carried out.

ELIGIBILITY:
Inclusion Criteria:

1. Type 2 diabetes mellitus newly-diagnosed (for group 1)
2. Type 2 diabetes and diabetic polyneuropathy (for group 2)
3. Availability of informed consent to participate in the study

Exclusion Criteria:

1. Refusal to sign informed consent to participate in the study
2. Presence of chronic diseases that require constant medication, except preparations for the correction of diabetes
3. Individual intolerance to the preparation
4. Infectious disease or fever during the period of inclusion
5. Refusal to take the preparation during the study
6. Non-compliance with inclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-10-03 (Actual); Primary Completion 2018-11-18 (Actual); Study Completion 2018-12-20 (Actual)

PRIMARY OUTCOMES:
Change in macrophages activation after single Cocarnit administration | 4 hours
  Measurement of serum-induced basal and stimulated by bacterial lipopolysaccharide secretion of TNF-alpha and basal and stimulated by IL-4 secretion of CCL-18 in primary cell culture of blood-derived monocytes-macrophages before and after 2 and 4 hours of Cocarnit administration. Changes are expressed in % of baseline secretion before the preparation administration.
Change in macrophages activation after 30-days Cocarnit administration | 30 days
  Measurement of serum-induced basal and stimulated by bacterial lipopolysaccharide secretion of TNF-alpha and basal and stimulated by IL-4 secretion of CCL-18 in primary cell culture of blood-derived monocytes-macrophages after 30 days of Cocarnit administration. Changes are expressed in % of baseline secretion before the preparation administration.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander N Orekhov, DSc, Prof, Principal Investigator — Institute for Atherosclerosis Research
Locations (1):
- Institute for Atherosclerosis Research, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shoelson SE, Lee J, Goldfine AB. Inflammation and insulin resistance. J Clin Invest. 2006 Jul;116(7):1793-801. doi: 10.1172/JCI29069. PMID 16823477
- [Background] Tilg H, Moschen AR. Inflammatory mechanisms in the regulation of insulin resistance. Mol Med. 2008 Mar-Apr;14(3-4):222-31. doi: 10.2119/2007-00119.Tilg. PMID 18235842
- [Background] Cave MC, Hurt RT, Frazier TH, Matheson PJ, Garrison RN, McClain CJ, McClave SA. Obesity, inflammation, and the potential application of pharmaconutrition. Nutr Clin Pract. 2008 Feb;23(1):16-34. doi: 10.1177/011542650802300116. PMID 18203961
- [Background] Gratchev A, Kzhyshkowska J, Kothe K, Muller-Molinet I, Kannookadan S, Utikal J, Goerdt S. Mphi1 and Mphi2 can be re-polarized by Th2 or Th1 cytokines, respectively, and respond to exogenous danger signals. Immunobiology. 2006;211(6-8):473-86. doi: 10.1016/j.imbio.2006.05.017. Epub 2006 Jul 21. PMID 16920487